## **BRITER Consent form**

**IRAS ID 216343** 

[Pick the date]



Patient Study Number:

## **CONSENT FORM**

## Title of Project: <u>B</u>rain <u>I</u>maging to predict <u>T</u>oxicity in <u>E</u>lderly patients after <u>R</u>adiotherapy (BRITER study)

Trial team: Dr C Lorimer, Dr J Brock, Dr L Welsh, Prof A Chalmers, Dr S Mills

| | | | Please initia | al all boxes |
|---|---|---|---|---|
| 1. | I confirm that I have read and understand the information sheet version | | | |
| 2. | . I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | 3. I understand that relevant sections of my medical notes, my scans and data collected during the study may be looked at by the trial team. I give permission for these individuals to have access to these records. | | | |
| 4. | I. I understand that my involvement will involve completing simple paper questionnaires and may involve undergoing an MRI scan with administration of a contrast agent through a cannula | | | |
| 5. | 5. I undertand that my GP will be informed that I am taking part in this study | | | |
| 6. | I agree to take part in the above st | udy. | | |
| Name of Participant | | Date | Signature | |
| | <u> </u> | | _ | |

Signature

Date

Consent form date of issue: 9.9.19 Consent form version number 4

Name of Trial team member